CLINICAL TRIAL: NCT06410911
Title: Analgesic Effect of Subcostal Transversus Abdominis Plane Block Versus Erector Spinae Block in Patients Undergoing Open Cholecystectomy Surgery
Brief Title: Subcostal Transversus Abdominis Block Versus Erector Spinae Block in Open Cholecystectomy
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mahmoud Abdellatif Mohamed, assistant lecturer of anaesthia an icu and pain managment, Sohag University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Soh-Med-24-04-01MD
Record Dates: First submitted 2024-05-03; First posted 2024-05-13 (Actual); Last update posted 2024-05-13 (Actual); Status verified 2024-05

CONDITIONS: Post Operative Pain, Acute
MeSH Terms: conditions — Pain, Postoperative

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Active Comparator): subcostal transversus abdominis plane block will be performed 50 patients undergoing open cholecystectomy surgery
  Interventions: Procedure: Subcostal Transversus Abdominis Plane block in patients undergoing open cholecystectomy surgery.; Drug: Sbcostal transversus Abdominis block and erector spinae block for both groups
- Group B (Active Comparator): Ultrasound-guided Erector spinae block will be performed 50 patients undergoing open cholecystectomy surgery
  Interventions: Procedure: Erector Spinae Block in patients undergoing open cholecystectomy; Drug: Sbcostal transversus Abdominis block and erector spinae block for both groups

INTERVENTIONS:
Procedure: Subcostal Transversus Abdominis Plane block in patients undergoing open cholecystectomy surgery. — Subcostal Transversus Abdominis Plain block will be performed under ultrasound guidance using a 5-10 MHz linear transducer. The needle will be inserted perpendicular to the skin 2 fingers below the costal
  margin, just lateral to the rectus abdominis muscle. After confirming the needle tip's location within the TAP, 20 mL of 0.25% bupivacaine will be injected on both sides in patients undergoing open cholicystectomy surgery.
  Arms: Group A
Procedure: Erector Spinae Block in patients undergoing open cholecystectomy — Ultrasound-guided Erector Spinae block using 20 mL of 0.25% bupivacaine will be injected bilaterally at the T7- T8 vertebral level in patients undergoing open cholecystectomy The probe will be advanced 3 cm to the right lateral direction and rotated 90 degrees, and the transverse processes will be determined . Next, 5 mL of 2% lidocaine will be administered to the predicted needle entry point. A 22-gauge, peripheral nerve block needle will cephalocaudally advanced by the in-plane technique. The needle tip will be continuously advanced toward the transverse process to 1-2 mm before contact with the transverse process. After negative aspiration, 20 ml of 0.25% bupivacaine will be injected with intermittent negative aspirations into the fascia of the erector spinae muscle.
  Arms: Group B
Drug: Sbcostal transversus Abdominis block and erector spinae block for both groups — Each patients group will recieve a type of block by injecting 20 ml of 0.25% bupivacaine on each side in patients undergoing open cholecystectomy

SUMMARY:
Open cholecystectomy is a surgical procedure involving the removal of the gallbladder through a traditional, open abdominal incision the surgeon makes an incision in the upper abdomen, exposes the gallbladder, and carefully disconnects and removes it. Postoperative pain management is a critical aspect of patient care following cholecytectomy surgery. Inadequate pain control can lead to a cascade of complications, including atelectasis, pneumonia, and delayed mobilization. These complications can prolong hospital stays, increase healthcare costs, and lead to patient dissatisfaction. Regional anesthesia techniques, such as subcostal transversus abdominis plane (TAP) block abd erector spinae block are commonly used to provide effective analgesia after cholecystectomy surgery. These techniques target the nerves that supply the surgical site, providing pain relief without the need for opioids. Opioids are associated with a number of side effects, including nausea, vomiting, constipation, and respiratory depression. Subcostal TAP block is a relatively new technique that has been shown to be effective in providing postoperative analgesia after upper abdominal surgery. This technique involves injecting local anesthetic into the TAP, a fascial plane that lies between the internal oblique and transversus abdominis muscles. The TAP block provides anesthesia to the nerves that supply the abdominal wall, including the subcostal nerves. Erector Spinae Plane Block is a newer technique targeting the dorsal rami of the T7-T12 spinal nerves, potentially offering broader analgesia encompassing the abdominal wall, thorax, and diaphragm. Early studies suggest improved pain control and respiratory function compared to traditional methods.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 65 years
* Both sex.
* American Society of Anesthesiologists (ASA) I-II Undergoing elective open cholecystectomy surgery.
* Patients who need at least 24hrs hospital admission.

Exclusion Criteria:

* Known allergy to local anesthetics
* Coagulopathy or bleeding disorders
* Severe respiratory disease
* Neurological disorders
* Pregnancy

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2024-06-01 (Estimated); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-07-01 (Estimated)

PRIMARY OUTCOMES:
Compare analgesic effect of both groups post open cholecystectomy surgery | 24 hours post operative
  to Compare the analgesic efficacy of subcostal transversus abdominis plain block and Erector Spinae block using Visual Analoug Score in both rest and coughing

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dai L, Ling X, Qian Y. Effect of Ultrasound-Guided Transversus Abdominis Plane Block Combined with Patient-Controlled Intravenous Analgesia on Postoperative Analgesia After Laparoscopic Cholecystectomy: a Double-Blind, Randomized Controlled Trial. J Gastrointest Surg. 2022 Dec;26(12):2542-2550. doi: 10.1007/s11605-022-05450-6. Epub 2022 Sep 13. PMID 36100826
- [Background] Viderman D, Aubakirova M, Abdildin YG. Erector Spinae Plane Block in Abdominal Surgery: A Meta-Analysis. Front Med (Lausanne). 2022 Feb 23;9:812531. doi: 10.3389/fmed.2022.812531. eCollection 2022. PMID 35280917